CLINICAL TRIAL: NCT07174960
Title: Life-Skills Training Program: Its Effect on Self-efficacy Among Patients With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdelmouttelb Abdelkawy, Assisstant lecturer, Master's degree, Psychiatric/Mental Health Nursing Faculty of Nursing Ain Shams University-Cairo-Egypt., Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NUR1. 25.01.527
Record Dates: First submitted 2025-08-21; First posted 2025-09-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders
Keywords: Life-Skills; Substance use disorders; self-efficacy; relapse; Addiction
MeSH Terms: conditions — Substance-Related Disorders; Recurrence; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: life-skills training program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quasi-experimental one group Pre-post test (Other): A 16-session program to boost self-efficacy & prevent relapse in SUD patients. It combines theoretical knowledge (5 sessions) with practical skills training (10 sessions) across cognitive skills, communication, and emotional skills. Uses interactive methods like role-play & discussion to teach vital life skills for recovery.
  Interventions: Behavioral: Life-Skills Training Program

INTERVENTIONS:
Behavioral: Life-Skills Training Program — This study aims to assess the impact of a life-skills training program on self-efficacy in patients with substance use disorders. The program is designed to prevent relapse by equipping individuals with crucial skills for managing triggers and challenges. It focuses on developing constructive coping strategies, effective stress and craving management techniques, social competencies like assertiveness, and emotional regulation abilities including anger control. By enhancing these domains, the intervention seeks to strengthen patients' confidence in their capacity to resist substance use and make adaptive decisions, thereby reducing relapse risk.

SUMMARY:
The goal of this clinical trial is to evaluate the effect of life-skills training program on self-efficacy among patients with substance in purposive sample male participants diagnosed with substance use disorders, aged from 20 :50 years old. Hypothesis Participants' Self-efficacy will be improved after implementation the life skills training program.

A quasi-experimental one-group pretest-post-test design was used

DETAILED DESCRIPTION:
1. Introduction and Rationale Substance Use Disorders (SUDs) represent a significant global public health challenge, characterized by a chronic, relapsing-remitting cycle influenced by biological, behavioral, and environmental factors. In Egypt, the prevalence is estimated at 5.9%, with the highest exposure among youth (15-25 years) and the highest treatment demand in the 25-35 age group. Alarmingly, relapse rates post-treatment can reach 40-75% within weeks to months, underscoring the inadequacy of detoxification-focused models that neglect psychosocial rehabilitation.

   A critical factor in sustaining recovery is self-efficacy (SE), particularly abstinence self-efficacy (ASE)-an individual's confidence in their ability to resist substance use in high-risk situations. Low SE is linked to poor motivation, increased withdrawal symptoms, and higher relapse susceptibility. Life skills, defined by the WHO as psychosocial competencies for adaptive and positive behavior, are foundational for managing triggers, stress, and social pressures. Training in these skills (e.g., problem-solving, communication, emotional regulation) is hypothesized to enhance SE, thereby reducing relapse risk. This study aimed to evaluate the effect of a structured life-skills training program on self-efficacy among patients with SUDs in a Cairo-based hospital.
2. Study Objectives and Hypothesis

   Primary Aim: To evaluate the effect of a life-skills training program on self-efficacy among patients with SUDs.

   Primary Hypothesis: Self-efficacy will significantly improve following the implementation of the life-skills training program.
3. Methods 3.1. Study Design: A quasi-experimental, one-group pre-test/post-test design was employed.

3.2. Setting: The study was conducted in the male addiction treatment and rehabilitation wards (detox and rehab) of the new building at El-Abbasia Mental Health Hospital in Cairo, Egypt.

3.3. Participants: A purposive sample of 45 male patients was recruited. Inclusion criteria were: age 20-50 years, a history of at least one relapse episode, being 3 weeks post-detoxification and engaged in rehabilitation, and being free from major comorbid physical (e.g., diabetes, hypertension) or psychiatric disorders. Sample size was determined via power analysis (α=0.05, β=0.15) based on a previous study.

3.4. Intervention (Life-Skills Training Program): The researcher-developed program, reviewed by supervisors and grounded in literature, comprised 15 core sessions (5 theoretical, 10 practical) plus orientation and closure sessions, delivered over 60 minutes each.

Theoretical Component (Sessions 1-5): Covered SUD concepts, substance classifications, risk factors, relapse triggers, recovery stages, craving management, and introductions to self-efficacy and life skills.

Practical Component (Sessions 6-15): Focused on applied skill-building across three domains:

Cognitive (Sessions 6-8): Problem-solving, decision-making, time management, and cognitive restructuring.

Communication (Sessions 9-12): Refusal, assertiveness, negotiation, and non-violent communication skills.

Emotional (Sessions 13-15): Anger management, meditation, relaxation techniques, and emotional regulation.

Pedagogy: Interactive methods were used, including open discussions, brainstorming, role-playing, demonstrations, videos, and handouts. Each session included homework review, feedback, objective setting, and a Q&A period.

3.5. Data Collection Tools:

Tool I: Interview Questionnaire: Collected socio-demographic and clinical data (substance type, history, treatment trials).

Tool II: Alcohol Abstinence Self-Efficacy Scale (AASE): A validated 40-item scale measuring confidence to abstain across four domains: Negative Affect, Social/Positive Situations, Physical Concerns, and Craving/Urges. Rated on a 5-point Likert scale (1=No Confidence to 5=Excellent Confidence). Total scores range from 40-200. Demonstrated high reliability in this study (Cronbach's α = 0.968).

3.6. Data Collection Procedure: The 7-month study (Feb-Aug 2024) followed stages: ethical approvals, baseline (pre-test) data collection using Tools I and II, program implementation for two cohorts (n=25, n=20), and post-intervention (post-test) data collection in September 2024 using the AASE.

3.7. Statistical Analysis: Data were analyzed using SPSS v26. Descriptive statistics (frequencies, percentages, means, standard deviations) described the sample. A paired t-test was used to compare pre- and post-intervention self-efficacy scores, with a significance level of p < 0.05.

Ethics: Approved by the Faculty of Nursing, Ain Shams University IRB (ID: NUR1.25.01.527). Informed consent was obtained from all participants

ELIGIBILITY:
Inclusion Criteria:

* male patients with substance use disorders
* aged 20 to 50 years
* who had experienced at least one relapse episode.
* All participants had completed a minimum of three weeks in detoxification and were actively involved in a structured rehabilitation program at the time of the study

Exclusion Criteria:

* Patients with chronic physical illnesses (e.g., diabetes, hypertension, or viral hepatitis)
* comorbid psychiatric disorders (e.g., schizophrenia, bipolar disorder, or depression) were excluded

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male (Substance use disorders are significantly more common among adult males, while prevalence among females remains very low. These patterns highlight notable gender disparities and underscore the predominance of substance use disorders in Egyptian adult men)
Enrollment: 45 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Interview Questionnaire | The assessment period for each participant was 10 weeks from the start of their participation in the study.
  Patients' characteristics. such as age, marital status (Single, Married, Divorced,& Widowed), Education levels (Read/ write, Primary, Secondary, and University or more) residence (Urban &Rural), Monthly income ( Enough, Fairly enough, & Not enough), Occupation (Don't work, Handicraft's work, and Administrative job) Number of Family members ( =2, =3, and ≥ 4)

SECONDARY OUTCOMES:
Clinical Data (Addiction History) | The assessment period for each participant was 10 weeks from the start of their participation in the study.
  Covered detailed information regarding the substance use history, including the types of substances used, duration of use (Less than 1 year, 1 -<5 years, 5 -<10 years, ≥ 10 years), route of administration (oral, inhalation, smoking, smell, and injection, history of previous treatment attempts (yse, no, number of times) types of treatment admissions (voluntary, & involuntary) and presence of substance cravings and numbers.

OTHER OUTCOMES:
Alcohol Abstinence Self-Efficacy Scale (AASE) | The assessment period for each participant was 10 weeks from the start of their participation in the study.
  The Alcohol Abstinence Self-Efficacy Scale (AASE; DiClemente et al., 1994) is a validated and previously published 40-item questionnaire assessing self-efficacy related to alcohol abstinence across four categories of high-risk situations every category includes 10 statements: negative affect, social/positive pressure, physical and other concerns, and withdrawal/urges. Participants rate their levels of temptation and confidence in each situation on a 5-point Likert scale such as each statement was rated on 5 points as Likert Skill Scale ranged by statistical from (1) No Confidence, (2) Low , (3) Moderate, (4) High, (5) Excellent and composite self-efficacy scores are calculated by subtracting temptation from confidence scores. The scale has demonstrated excellent internal consistency (Spearman-Brown r =.95), and in this study, the adapted translated version for substance abstinence showed high reliability (Cronbach's alpha = 0.912) validated by the researchers

CONTACTS AND LOCATIONS:
Overall Officials: Abdelmouttelb Ab Abdelkawy, Ass/Lecturer, Principal Investigator — Psychiatric/Mental Health Nursing Faculty of Nursing Ain Shams University-Cairo-Egypt.; Fatma Mo Ibrahim, Assist/Prof, Study Director — Psychiatric/Mental Health Nursing , Faculty of Nursing Ain Shams University-Cairo-Egypt.; Fatma At Abdelsalhen, Assist/Prof, Study Director — Psychiatric/Mental Health Nursing , Faculty of Nursing Ain Shams University-Cairo-Egypt.; Sahar Ma Elewa, Professor, Study Chair — Psychiatric/Mental Health Nursing Faculty of Nursing Ain Shams University-Cairo-Egypt.
Locations (2):
- Egypt (2):
  - El Abbasia Mental Health Hospital, Cairo, El Abbasia
  - faculty of Nursing Ain Shams University, Cairo, El Abbasia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Informed Consent Form (ICF), all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: present

REFERENCES:
- [Background] Moshki M, Hassanzade T, Taymoori P. Effect of Life Skills Training on Drug Abuse Preventive Behaviors among University Students. Int J Prev Med. 2014 May;5(5):577-83. PMID 24932389
- [Background] Ebrahem SM, Badawy SA, Hassan RA, Radwan HA, Shokr EA, Hussein AA. Effect of Telehealth Nursing Intervention on Psychological Status and Coping Strategies Among Parents During COVID-19 Pandemic. Holist Nurs Pract. 2023 Jan-Feb 01;37(1):34-44. doi: 10.1097/HNP.0000000000000561. PMID 36378090
- [Result] Abdelmouttelb AA, Elewa SMM, Abdelsalhen FA, Ibrahim FM. Life-skills training program: its effect on self-efficacy among patients with substance use disorders. BMC Psychol. 2026 Jan 21;14(1):119. doi: 10.1186/s40359-025-03907-2. PMID 41566382

DOCUMENTS (2):
  • Study Protocol (2023-04-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT07174960/Prot_000.pdf
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT07174960/ICF_001.pdf